CLINICAL TRIAL: NCT05702515
Title: Vascular Positioning System G4 Algorithm ECG Data Collection for Model Training Study, A Single Center Prospective Clinical Study
Brief Title: Vascular Positioning System G4 Algorithm ECG Data Collection for Model Training Study
Status: Completed | Type: Observational
Sponsor: Teleflex (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-03
Record Dates: First submitted 2023-01-17; First posted 2023-01-27 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-02

CONDITIONS: Peripheral ICC
Keywords: VPS; VPS G4; Vascular Positioning System G4; PICC navigation and tip confirmation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult male patients scheduled to receive a PICC insertion: Adult male patients scheduled to receive a PICC insertion using the Vascular Positioning System G4 tip navigation system
  Interventions: Other: Digital ECG Data Collection

INTERVENTIONS:
Other: Digital ECG Data Collection — synchronized digital data collected from the G4 and ECG machines during the PICC insertion procedure

SUMMARY:
The objective of this study is to collect intravascular and extravascular echocardiogram (ECG) data from subjects receiving peripherally inserted central catheters (PICC) while using the Vascular Positioning System G4 and a 12 lead ECG machine. The data obtained will be used to update the G4 algorithm.

DETAILED DESCRIPTION:
This study seeks to collect synchronized digital data collected from the G4 and ECG machines during the PICC insertion procedure. A copy of the data will be downloaded from the G4 and ECG machines and submitted to the sponsor. Both the G4 and the ECG machine used for data collection in this study are FDA cleared/approved.

Study Design: This is a single center prospective clinical study. All enrolled subjects will receive a 12-lead ECG during PICC insertion and a chest x-ray post insertion. ECG lead will be documented via photographic imaging.

Duration of Subject Study Participation: Each subject's participation will start at the time of signing the informed consent and terminate upon completion of the x-ray.

ELIGIBILITY:
Inclusion Criteria:

* Male

  * 21 years of age or older
  * Scheduled for PICC insertion using the VPS G4 system
  * Willing to allow thoracic photos to be obtained after ECG lead placement

Exclusion Criteria:

* Female

  * ˂ 21 years of age
  * Patient has a pacemaker
  * Patient condition precluding ECG use and lead placement
  * Patient condition precluding radiographic imaging
  * Unwilling to allow thoracic photos to be obtained after ECG lead placement

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male subject over the age of 21
Study Population: Adult male patients scheduled to receive a PICC insertion using the G4 tip navigation system may be considered for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Puga, B.S.B., Study Director — Teleflex Inc; Deborah H Allen, PhD, Principal Investigator — Duke University; Britt M Meyer, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data collected simultaneously from the G4 system and a 12-lead ECG machine during PICC insertion in adult subjects will be used for refining the next generation G4 algorithm model.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Willing adult patients scheduled to receive a PICC insertion using the G4 tip navigation system were screened and enrolled in the study.
Groups:
- Adult Patients Scheduled to Receive a PICC Insertion: Adult patients scheduled to receive a PICC insertion using the Vascular Positioning System G4 tip navigation system
  Digital ECG Data Collection: synchronized digital data collected from the G4 and ECG machines during the PICC insertion procedure
Period: Overall Study
Arm/Group | Adult Patients Scheduled to Receive a PICC Insertion
Started | 27
Completed | 20
Not Completed | 7
Not completed — 7 patients were excluded due to the inability to complete a chest radiograph. | 7

BASELINE CHARACTERISTICS:
Population: Adult patients scheduled to receive a PICC insertion using the G4 tip navigation system and completed a chest x-ray were enrolled in the study.
Arm/Group | Adult Patients Scheduled to Receive a PICC Insertion
Number analyzed (Participants) | 20
Age, Customized [Number; unit: participants who completed chest xray] — Age 22 years old and older
  participants who completed chest xray
    Subject 22 years old or older scheduled to receive a PICC using the VPS G4 and completion of xray | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: VPS G4 System Digital Data vs GE MAC 5500 Ecg Machine Data
Description: All subjects for this study had their ECG recorded by the VPS G4 and GE MAC 5500 simultaneously. VPS G4 digital captured data recorded at 11.667 MHz measuring ISPTA.3 (mW/cm2) vs Digitally captured data from the GE MAC 5500 ECG Machine at a sample resolution of 4.88 μV/LSB @ 250 sps, 1.22 μV/LSB @ 500 sps and a frequency response of -3 dB @ 0.01 to 150 Hz vs time (s).
Time Frame: From time of consent through completion of chest x-ray
Measure: Number; unit: subjects who digital data was captured
Arm/Group | Adult Patients Scheduled to Receive a PICC Insertion
Number analyzed (Participants) | 20
subjects who digital data was captured | 20

ADVERSE EVENTS:
Time Frame: Study conducted between June 2023- July 2024. Subjects were evaluated from the time they were consented through completion of the chest x-ray.
Description: Number of AE Number of SAE Number of UADE 0 0 0
  There were no reported AE/SAE/UADE reported during this study due to the short nature of the study. The average time from consent to completion of the study was usually less than 3 hours.
Groups:
- Adult Patients Scheduled to Receive a PICC Insertion: This was a single arm study evaluating consenting adult patients scheduled to receive a PICC insertion using the Vascular Positioning System G4 tip navigation system being enrolled and evaluated. Digital ECG Data Collection, synchronized digital data collected from the G4 and ECG machines during the PICC insertion procedure, was collected for all subjects enrolled.
Arm/Group | Adult Patients Scheduled to Receive a PICC Insertion
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/15/NCT05702515/Prot_SAP_000.pdf